CLINICAL TRIAL: NCT01048931
Title: To Compare to Single-port Access Laparoscopic-assisted Vaginal Hysterectomy (LAVH) and Multiple Ports LAVH: A Randomized Controlled Trial
Brief Title: Single-port Access Laparoscopic-assisted Vaginal Hysterectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Chen-Hsen Lee, MD, Chairman, Taipei Veterans General Hospital,Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB 98-10-03
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Uterine Myomas; Adenomyosis
Keywords: Single-port, laparoscopic-assisted, vaginal hysterectomy
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-port LAVH (Experimental): single port LAVH
  Interventions: Procedure: single-port LAVH

INTERVENTIONS:
Procedure: single-port LAVH — single-port LAVH

SUMMARY:
Minimally invasive surgery has become the standard treatment for many gynecologic disease processes. In the last decade, numerous studies have demonstrated that laparoscopic approaches to various gynecologic oncology conditions-particularly for early-stage endometrial and cervical cancers as well as select pelvic masses-is feasible and results in shorter hospital stays, improved quality of life and comparable surgical and oncologic outcomes to abdominal staging [1-5].For instance, the typical gynecologic robotic surgical procedure will require Two to three 5-mm ports and one 12-mm laparoscopic ports. Recently, an even less invasive alternative to conventional laparoscopy surgery has been developed: laparoendoscopic single-site surgery (LESS), also known as single-port surgery. Single port laparoscopy is an attempt to further enhance the cosmetic benefits of minimally invasive surgery while minimizing the potential morbidity associated with multiple incisions. However, to our knowledge, there are no randomize control trial to evaluate of single port or multiple ports laparoscopic surgery in gynecologic disorders. The purpose of this study was to assess the feasibility of SPA-LAVH in the treatment of benign uterine disease.

DETAILED DESCRIPTION:
Overall Study Design:

Participants:

This clinical controlled trial will be undertaken among patients who will receive laparoscopic-assisted vaginal hysterectomy.

Interventions:

All the patients will receive laparoscopic surgery using CO2 gas as distension medium. At the end of the surgery, in the control group, CO2 was removed by passive exsufflation through the port site. The patients will be placed in the Trendelenburg position (30 degrees).

In the intervention group: 50 patients receive the single port-access laparoscopic-assisted vaginal hysterectomy. Under general anesthesia, the patient was positioned in the supine position with the legs extended, and prepped and draped in the routine sterile fashion. The legs were protected with foam padding. At the start of surgery, a 2-cm intraumbilical incision was made. Adhesiolysis was performed if adhesions between the viscera and peritoneum existed from prior abdominal surgery or past abdominopelvic infection. The single-port system was made based on a modification of Lee et al. procedure [8]. After insertion of the wound protractor (Alexis X-small for 2-4 cm incisions, Applied Medical, CA, USA) into the abdominal cavity, the extraabdominal portion of the wound protractor was rolled up with the wrist portion of a surgical glove (TriflexLP, 7-0; Cardinal Health, OH, USA; Fig. 1). The finger portion of the glove was resected and tied to prevent leakage of carbon dioxide. The first trocar sleeve for laparoscopy was created after a small incision in the upper portion of the glove was made in the midline. After insertion of a trocar sleeve, the surrounding glove was lifted up with two mosquito forceps and tied to the trocar sleeve. Next, carbon dioxide was insufflated to maintain intra-abdominal pressure at 12-14 mmHg, depending on age and condition of the patient. Five- or 10-mm laparoscopes were used as needed. These laparoscopes have an incorporated light source within the camera head that does not compete for the very limited space in the port site. One or two additional 5-mm trocar sleeves were introduced through the single port system to make an imaginary triangle with the previous port for the camera to avoid clashing and to maximize surgical movement. A uterine manipulator was inserted to optimize visualization and accessibility in the surgical field . Then the laparoscopic assisted vaginal hysterectomy was perform as usual. Finally, the approach to the fascia and peritoneum is easier via the umbilicus than an extra-umbilical area; the peritoneum and fascia were approximated and closed layer by layer with 2-0 Vicryl suture and the skin was selectively sutured .

In the control group: 50 patients receive the multiple ports-access laparoscopic-assisted vaginal hysterectomy (traditional LAVH, usually 3-4 ports) as previous described.

Objectives and outcomes:

The main objective of this trial is to assess the efficacy and safety of single port-access laparoscopic-assisted vaginal hysterectomy. The operative time, weight of the uterus, blood loss and hospital stay will be record, respectively. The pain score is based on the visual analogue scale in which patients record the intensity of their pain 12, 24, and 48 hours after surgery. The rate of multiple ports laparoscopy convert to transabdominal hysterectomy will be record. The rate of single ports laparoscopy convert to multiple ports laparoscopy or transabdominal hysterectomy will be record.

The morbidity (wound infection, hernia, fever...) associated with surgery will be noted, too.

Randomization process:

Treatment allocation was performed in accordance with a computer-generated randomization sequence using numbered, sealed envelopes.

Main Inclusion/ Exclusion Criteria Inclusion

1. Patients receive laparoscopic-assisted vaginal hysterectomy (LAVH)
2. American Society of Anesthesiologists (ASA) physical status of patient: classification I-II

Exclusion

1. The procedure will be required to conversion to laparotomy.
2. Any cardio-vascular diseases.
3. Malignant disease

Number of subjects: 100 Methods: In the intervention group : 50 patients receive the single port-access laparoscopic-assisted vaginal hysterectomy.

In the control group : 50 patients receive the multiple ports-access laparoscopic-assisted vaginal hysterectomy (traditional LAVH, usually 3-4 ports).

Planned Study Timelines:

(submission date to Health authority in 1st country, dates of start and end of subject enrolment, end of study) Dates of start: Aug., 2009 End of study: Aug., 2011

Evaluation of efficacy:

Sample size:

In calculating the sample size required, the primary assessment was the post-operative time and blood loss. We determined a required sample size of 50 patients per group for a two-tailed X2 test with 80% power and a P level of .05. Thus a total of 100 analyzable patients were obtained for this study.

Endpoints:

We will follow the patients until one month after the surgery. The primary outcome measure of this trial is the effect and safety of single port-access laparoscopic-assisted vaginal hysterectomy.

Statistical analysis plan:

Normality was assessed by means of the Kolmogorov-Smirnov test. Differences between the groups were analyzed by using an unpaired two-tailed t test for continuous variables and the X2 test for binomial outcomes (Stata 10 Edition for Windows, StataCorp LP, College Station, TX). The pain scores over time and their interaction with the intervention were analyzed by means of the analysis of variance for repeated measures (SPSS 15.0.0, SPSS Inc., Chicago, IL). Effects were considered statistically significant for P<.05

ELIGIBILITY:
Inclusion Criteria:

* Patients receive laparoscopic-assisted vaginal hysterectomy (LAVH)
* American Society of Anesthesiologists (ASA) physical status of patient: classification I-II

Exclusion Criteria:

* The procedure will be required to conversion to laparotomy.
* Cancer

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy and safety of single port-access laparoscopic-assisted vaginal hysterectomy. The pain score and morbidity associated with surgery will be noted. | 1 year

SECONDARY OUTCOMES:
To evaluate the cosmetic outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, MD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Veterans General Hospital -Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Lee YY, Kim TJ, Kim CJ, Kang H, Choi CH, Lee JW, Kim BG, Lee JH, Bae DS. Single-port access laparoscopic-assisted vaginal hysterectomy: a novel method with a wound retractor and a glove. J Minim Invasive Gynecol. 2009 Jul-Aug;16(4):450-3. doi: 10.1016/j.jmig.2009.03.022. Epub 2009 May 31. PMID 19487164
- [Derived] Chen YJ, Wang PH, Ocampo EJ, Twu NF, Yen MS, Chao KC. Single-port compared with conventional laparoscopic-assisted vaginal hysterectomy: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):906-912. doi: 10.1097/AOG.0b013e31820c666a. PMID 21422864